CLINICAL TRIAL: NCT03828487
Title: Performance Comparison of Masimo O3 Regional Oximetry Sensors in Neonates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated study due to project timeline.
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RAMA0004
Record Dates: First submitted 2019-01-10; First posted 2019-02-04 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Regional Saturation of Oxygen (rSO2)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neonatal Test group (Experimental): Subjects will receive a Masimo O3 Neonatal sensors as well as a 510(k) cleared sensor.
  Interventions: Device: Masimo O3 Neonatal Sensors; Device: 510(k) cleared sensor

INTERVENTIONS:
Device: Masimo O3 Neonatal Sensors — Regional Oximetry sensor for Neonates
Device: 510(k) cleared sensor — Cleared Regional Oximetry sensor for Neonates

SUMMARY:
The aim of the study is to compare the performance of the O3 cerebral oximeter and sensor to a 510(k) cleared NIRS (Near-Infrared Spectroscopy) device on neonatal subjects based on data collected from the cutaneously placed forehead sensors. Due to the design of the systems, the devices will be used serially instead of concurrently. Because of this timing, changes in patient state may not be reflected in measurements collected by both devices.

ELIGIBILITY:
Inclusion Criteria:

* Less than 10 kg
* Subjects less than or equal to 28 days old

Exclusion Criteria:

* Underdeveloped skin at sites of sensor placement
* Jaundice or bilirubin levels out of normal range
* Subject has skin abnormalities affecting the sensor placement area such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, or substantial skin breakdown that would prevent monitoring of oxygenation levels during the study
* Subject deemed not eligible based on Principal Investigator's judgment

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neonatal Test Group
Started | 8
Completed | 7
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neonatal Test Group
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With rSO2 Collected
Description: In order to obtain the RMS value, rSO2 values collected from the control device (510(k) cleared regional oximetry sensor) is subtracted from the rSO2 values collected from the investigational device (Masimo O3 neonatal sensors) for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the RMS Error value.
Time Frame: Data collection period; alternating sensors every 5 minutes for up to 20 minutes.
Population: Study was prematurely terminated. Study did not reach the target number of subjects needed to achieve minimum sample size determination and was insufficient to produce statistically reliable results.
Measure: Count of Participants; unit: Participants
Arm/Group | Neonatal Test Group
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Neonatal Test Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Study did not reach the target number of subjects needed to achieve minimum sample size determination and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03828487/Prot_SAP_000.pdf